CLINICAL TRIAL: NCT03001947
Title: IgA Nephropathy Registration Initiative of High Quality (INSIGHT)
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Professor, Sun Yat-sen University
Other Study IDs: INSIGHT
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: IgA Nephropathy
Keywords: IgA nephropathy; All-cause mortality; Cardiovascular mortality; A composite renal outcome
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — The serum, urine, DNA and renal tissue will be collected.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- IgAN patients: Biopsy-proven primary IgAN patients
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Registration of all IgAN patients in the First Affiliated Hospital of Sun Yat-sen University and other hospitals which have signed the contract in China.

SUMMARY:
The investigators are registering all biopsy-proven primary IgA nephropathy (IgAN) patients at recruited hospitals and developing a IgAN database in China. Patients will be follow-up every one year, and both baseline and follow-up information will be entered into the registration system. All-cause and cardiovascular mortality and a composite renal outcome of doubling of serum creatinine and end stage renal failure (ESRD, defined as initiation of dialysis or kidney transplantation) of IgAN patients will be compared using the IgAN database.

DETAILED DESCRIPTION:
The investigators are registering all biopsy-proven primary IgA nephropathy (IgAN) patients, and developing a IgAN database in China. Patients' demographic characteristics (including age, gender, height, weight, BMI, smoking, drinking, and education), clinical characteristics (including systolic blood pressure, diastolic blood pressure, primary cause of ESRD, and lab measurements of serum and urine), complications, drug information at the baseline will be collected. Patients will be follow-up every one year, the demographic and clinical characteristics, complications and drug information of patients will be collected at each visit. The investigators also record the clinical events at each visit, such as mortality (including all-cause mortality and cardiovascular disease mortality), ESRD (defined as initiation of dialysis or kidney transplantation) and hospitalization for any cause. All-cause and cardiovascular mortality and a composite renal outcome of doubling of serum creatinine and ESRD for IgAN patients will be compared using the IgAN database.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven primary IgAN patients;
2. age ≥14 years old
3. Adequate biopsy sample containing ≥8 glomeruli.

Exclusion Criteria:

Secondary causes of mesangial IgA deposition, such as Henoch-Schonlein purpura nephritis, systemic lupus erythematosus, liver cirrhosis and et al; eGFR≤15ml/min/1.73m2 at biopsy.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Biopsy-proven primary IgAN patients
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2012-11; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
All-cause and cardiovascular mortality of IgAN patients | 10 years
A composite renal outcome of IgAN patients | 10 years
  The composite renal outcome defined as doubling of serum creatinine and ESRD (defined as initiation of dialysis or kidney transplantation).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes